CLINICAL TRIAL: NCT03735563
Title: Premedication for Less Invasive Surfactant Administration
Acronym: LISA-Med
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oulu (Other)
Collaborators: Oulu University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OY062018
Record Dates: First submitted 2018-11-07; First posted 2018-11-08 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Surfactant Deficiency Syndrome Neonatal
Keywords: less invasive surfactant administration; premedication
MeSH Terms: conditions — Pulmonary Atelectasis | interventions — Ketamine; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The investigators and medical staff are blinded to the fact which study medication is given. A pharmacist or a nurse not participating in treatment of the child in question prepares the drug. Preparation of the study drug is done in a different location than where the treatment takes place.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketamine (Experimental): Individuals needing the LISA will receive premedication as follows: caffeine (in case of gestational age <32 weeks and not already given), glycopyrrolate, and randomly either ketamine or fentanyl.
  Interventions: Drug: Ketamine
- Fentanyl (Experimental): Individuals needing the LISA will receive premedication as follows: caffeine (in case of gestational age <32 weeks and not already given), glycopyrrolate, and randomly either ketamine or fentanyl.
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Ketamine — Individuals will receive randomly either ketamine or fentanyl as a premedication
  Other Names: Ketanest-S
  Arms: Ketamine
Drug: Fentanyl — Individuals will receive randomly either ketamine or fentanyl as a premedication
  Other Names: Fentanyl-Hamel
  Arms: Fentanyl

SUMMARY:
Early respiratory management of preterm infants immediately after birth should be as gentle as possible. With this so-called developmental approach, unnecessary invasive methods can be avoided or at least postponed. This kind of "soft landing" allows cardiorespiratory transition with fewer adverse outcomes. Less invasive surfactant administration (LISA) is a technique that involves delivery of surfactant to a spontaneously breathing infant through a thin catheter. This technique minimizes the risk for neonatal lung injury caused by positive pressure ventilation. LISA is nowadays widely used in neonatal intensive care units (NICU). Although less invasive, newborns exposed to this procedure need premedication prior the procedure. There is no consensus, which drug would be the optimal premedication for LISA and the research on this topic is lacking. An ideal premedication would treat the procedural pain without suppressing the infant's own breathing. The sedation and analgesia should start fast but the effect should be short-acting with as few adverse effects as possible. The aim of this randomized, controlled trial (RCT) is to evaluate the feasibility, efficacy and safety of LISA protocol with the premedication of either ketamine or fentanyl by investigating whether one or the other is associated with lower rate of adverse events, hence would be preferred choice for premedication protocol.

DETAILED DESCRIPTION:
All infants fulfilling the inclusion criteria during the study period are asked to participate in this randomized controlled trial of LISA premedication. Written informed parental consent is acquired from all of the participants. After the consent, individuals needing the LISA will receive premedication as follows: caffeine (in case of gestational age <32 weeks and not already given), glycopyrrolate, and randomly either ketamine or fentanyl. The investigators and medical staff are blinded to the fact which study medication is given. This study is a pilot study and 20 patients are recruited for both groups. Randomization is done in the blocks of four.

S-ketamine (Ketanest-S 5 mg/ml) or fentanyl (Fentanyl-Hamel diluted to 5 μg/ml) is used as a masked study drug. Both study drug solutions appear equally transparent. Drug administration is started with glucopyrrolate (Robinul 0.2 mg/ml), which is given intravenously at a dose of 5 µg/kg. Thereafter, the masked study drug is administered intravenously slowly in one to two minute injection of 0.2 ml/kg. In this way, doses of S-ketamine 1 mg/kg or alternatively fentanyl 1 μg/kg is received. After five minutes (from the beginning of administration of the study drug), videolaryngoscopy is started. If the study drug does not have sufficient effect, the study drug may be repeated with the same dose. If study drug fails to give appropriate conditions to LISA procedure, midazolam 0,1 mg/kg can be used as an additional drug.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age at birth ≥26 weeks
* Respiratory insufficiency managed with non-invasive respiratory support (nasal continuous positive airway pressure or high-flow)
* Requirement for oxygen to maintain oxygen saturation in the target range and need for surfactant treatment (according to clinician's assessment)
* If further doses of surfactant are needed, patient can be re-randomized

Exclusion Criteria:

* Severe RDS with high oxygen requirements, severe respiratory acidosis and/or widespread atelectasis radiologically, such that ongoing ventilator support will be necessary after surfactant therapy (intubation in preferable to LISA if FiO2 >40% at GA <28 weeks and >60% at GA ≥28 weeks)
* Maxillo-facial, tracheal or known pulmonary malformations
* Any known chromosomal abnormality or severe malformation
* An alternative cause for respiratory distress (e.g. congenital pneumonia or pulmonary hypoplasia)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-02-11 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Adverse event | 1 hour
  The need of positive pressure ventilation (PPV), intubation, heart rate below 80 per minute, mean arterial pressure change more than 20%, pH change more than 0.4, and CO2 change more than 20%, and saturation <85 for more than 1 minute

SECONDARY OUTCOMES:
Duration of the procedure | 1 hour
  Duration of the procedure is evaluated retrospectively from the recording of the videolaryngoscopy (an attempt begins when the laryngoscope enters the mouth and ends with LISACath in the trachea)
Number of attempts to get the catether intratracheally | 1 hour
  Number of attempts to get the catether intratracheally is evaluated retrospectively from the recording of the videolaryngoscopy (one laryngoscopy = one attempt)
Pain score NIAPAS | 1 hour
  Pain will be scored with validated Neonatal Infant Acute Pain Assessment Scale (NIAPAS) tool. The scale includes five behavioral and three physiological indicators, and takes into account the gestational age of neonates as a contextual factor. The indicators are rated on a 2, 3, or 4-point scale for a possible total score of 18. Assessments of each neonate include alertness, facial expressions, crying, muscle tension, reaction to handling, and breathing. In addition, the neonates on monitors are assessed for changes in heart rate and oxygen saturation (Copyright Pölkki T, Korhonen A, Axelin A. 2013)
The need for additional dosing of study drug or midazolam (number of addtional dosages) | 1 hour
  If the study drug does not have sufficient effect, the study drug may be repeated with the same dose. If study drug fails to give appropriate conditions to LISA procedure, midazolam 0,1 mg/kg can be used as an additional drug.
Edi-signals | 1 hour
  Special Edi (Electronic Diaphragm Monitoring) Catheter is placed to read the electrical activity of the diaphragm. Edi min and Edi max in different time points will be collected.

CONTACTS AND LOCATIONS:
Overall Officials: Riitta Marttila, MD, docent, Principal Investigator — Oulu University and Oulu University Hospital
Locations (1):
- Oulu University Hospital, Oulu, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sweet DG, Carnielli V, Greisen G, Hallman M, Ozek E, Plavka R, Saugstad OD, Simeoni U, Speer CP, Vento M, Visser GH, Halliday HL. European Consensus Guidelines on the Management of Respiratory Distress Syndrome - 2016 Update. Neonatology. 2017;111(2):107-125. doi: 10.1159/000448985. Epub 2016 Sep 21. PMID 27649091
- [Background] Vento M, Dargaville P, Bohlin K, Herting E & Roehr C LISA Training Advisory Board Report.
- [Background] Polkki T, Korhonen A, Axelin A, Saarela T, Laukkala H. Development and preliminary validation of the Neonatal Infant Acute Pain Assessment Scale (NIAPAS). Int J Nurs Stud. 2014 Dec;51(12):1585-94. doi: 10.1016/j.ijnurstu.2014.04.001. Epub 2014 Apr 18. PMID 24815773